CLINICAL TRIAL: NCT05596097
Title: Clinical Research for Efficacy and Safety of Zanubrutinib in Maintenance Therapy of DLBCL Patients With Initial Remission
Brief Title: Zanubrutinib in Maintenance Therapy of DLBCL Patients With Initial Remission
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LanZhou University (Other)
Collaborators: BeOne Medicines (Industry)
Responsible Party: Principal Investigator, Bei Liu, Chief Physician, Clinical Professor，Deputy Director of Hematology Department, LanZhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEBUBU22
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL)
Keywords: Diffuse Large B-cell Lymphoma (DLBCL); Maintenance Therapy; Zanubrutinib; Rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib

STUDY DESIGN:
Intervention Model Description: According to the initial treatment plan of the patients, the patients were divided into R-CHOP and R-chemo groups. Both groups received zanubrutinib maintenance therapy after induction and consolidation therapy reached the maximum curative effect. With event-free survival (EFS) as the primary endpoint, partial remission (PR) to CR conversion rate, progression-free survival (PFS), and overall survival (OS) as secondary endpoints, adverse events (AEs) were assessed. ) incidence and related mechanisms during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): According to the initial treatment plan of the patients, the patients were divided into R-CHOP and R-chemo groups. Both groups received zanubrutinib 160 mg bid p.o. d1-28 maintenance treatment for 12 months after induction and consolidation therapy reached the maximum efficacy.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib, 180mg, bid, p.o., d1-28; Treatment cycles every 28 days

SUMMARY:
This trial is a single-center, single-arm, prospective clinical study to investigate the efficacy and safety of zanubrutinib maintenance therapy in patients with diffuse large B-cell lymphoma (DLBCL) in Initial remission. The patients were divided into two categories: 1) Zanubrutinib maintenance therapy was started after R-CHOP induction and consolidation therapy reached maximum efficacy; 2) Initiate zanubrutinib maintenance therapy after maximal response to induction and consolidation therapy with or without rituximab (R-chemo). Therefore, the data in this study will reflect the efficacy and safety of zanubrutinib in the maintenance treatment of DLBCL patients with initial remission, and will provide new insights into the clinical application of zanubrutinib.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most common aggressive malignant lymphoma, and because it is sensitive to chemotherapy, approximately 50% to 70% of patients can achieve a cure after first-line treatment. However, in recent years, it has been found that more than 30% of patients experience relapse within two years after first-line treatment, which is a serious health threat and requires urgent secondary treatment. To reduce the recurrence of DLBCL and improve the survival rate of patients, clinical researchers have long been dedicated to the maintenance treatment of DLBCL patients after first-line treatment, aiming to kill tumor cells and reduce the risk of recurrence through continuous drug administration, thus enabling patients to survive with the tumor for a long time. Several clinical trials are currently underway with rituximab, ibrutinib, lenalidomide, and thalidomide, but safer and more effective maintenance regimens have yet to be identified.

Zanubrutinib, a new-generation BTK inhibitor, is the first anti-tumor drug developed locally in China and approved for marketing in the US. Zanubrutinib inhibits the activation of the BCR signaling pathway by specifically binding to cysteine residues at the active site of BTK to form a covalent bond that irreversibly inactivates them, thereby inhibiting BTK and improving the tumor microenvironment, inhibiting malignant proliferation and inducing apoptosis in tumor B cells. Several clinical studies have demonstrated that ibrutinib alone and in combination is no less effective than ibrutinib in the treatment of DLBCL, and has a better safety and tolerability profile.

This study proposes to use Zanubrutinib for maintenance treatment in DLBCL patients in remission after primary treatment and to evaluate the efficacy and safety of patients to provide new insights into the clinical use of Zanubrutinib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with DLBCL who are diagnosed according to the 2021 NCCN Guidelines for B-cell Lymphoma, aged ≥18 years;
2. Don't received treatment;
3. Measurable lesions: at least 1 lymph node lesion > 1.5 cm in longest dimension, or at least 1 extranodal lesion > 1.0 cm in longest dimension, and at least 2 measurable lesions accurately measured vertical diameter;
4. Clinical stage II (not suitable for local radiotherapy), III, IV (Ann Arbor stage); Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
5. Intermediate-high-risk /high-risk group: International Prognostic Index (IPI) score 3-5, aa-IPI score 2-3 or NCCN-IPI score ≥4;
6. Expression of MYC, BCL-2 and BCL-6 (detected by immunohistochemistry, qualitative or quantitative detection), or MYD88, CD79A/CD79B [9] and TP53 genetic abnormality [10];
7. Patients with non-bone marrow invasion:

   1. The absolute value of neutrophils≥1.5×109/L
   2. Platelets ≥100×109/L (judged by the investigator according to the condition, the minimum can be ≥75×109/L)
   3. Hemoglobin ≥ 90g/L;

9. The level of biochemical indicators meets the following requirements:

1. Renal function: endogenous creatinine clearance rate > 30ml/min;
2. Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal range (ULN); total bilirubin ≤ 2 × ULN (unless Gilbert syndrome is diagnosed);
3. Coagulation function: international normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.5×ULN; 9. life expectancy ≥ 3 months; 10. The patient and family members agree and sign an informed consent form.

Exclusion Criteria:

1. Lymphoma with central nervous system invasion or mediastinal large B-cell lymphoma, diagnosis or treatment of malignant tumors other than DLBCL;
2. Cannot tolerate zanubrutinib treatment, or have hypersensitivity reactions to any components of the study drug;
3. Significant cardiovascular disease, including:

   1. Myocardial infarction within 6 months prior to screening;
   2. Unstable angina pectoris occurring within 3 months prior to screening;
   3. Clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes);
   4. QTc (corrected by Fridericia formula): >450ms in men, >470ms in women, or other ECG abnormalities, including history of second-degree type II atrioventricular (AV) block or third-degree AV block;
   5. Any grade 3 or 4 heart disease as defined by the New York Heart Association (NYHA) functional class;
   6. Echocardiography (ECHO) showing left ventricular ejection fraction (LVEF) ≤40% (AHA, 2022);
   7. Uncontrolled hypertension at screening, manifested as systolic blood pressure ≥180 mmHg and diastolic blood pressure ≥110 mmHg on at least two consecutive blood pressure measurements;
4. Requires continuous treatment with strong or moderate CYP3A inhibitors/inducers. Patients are not eligible if they have taken strong or moderate CYP3A inhibitors/inducers within 7 days prior to the first dose of study drug (or have taken these drugs for less than 5 half-lives);
5. Hepatitis B virus (HBV-DNA) ≥ 1x10^3 copies/mL or HBV-DNA > 200 IU/mL or active hepatitis C virus (HCV), or human immunodeficiency virus (HIV) Serologically positive;
6. Obvious bleeding tendency, such as a history of stroke, intracranial hemorrhage within 6 months, or a history of surgery within 4 weeks;
7. Serious infectious diseases at the same time;
8. Refuse to take reliable contraceptive methods during pregnancy, lactation or appropriate age;
9. Participate in another clinical trial of lymphoma treatment at the same time;
10. Unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | up to 36 months
  EFS was defined as the time from initiation of zanubrutinib maintenance therapy to the occurrence of any event, including death, disease progression, change in chemotherapy regimen, change to chemotherapy, addition of other treatments, occurrence of fatal or intolerable side effects, etc. Whichever occurs first.

SECONDARY OUTCOMES:
Conversion rate of partial response (PR) to CR | up to 36 months
  the total proportion of patients who had a partial response to initial therapy converted to CR at any time point after starting zanubrutinib maintenance therapy and will be reported as converted to CR at 3, 6, 12 months, and any other time point.
Progression-free survival (PFS) | up to 36 months
  PFS was defined as the duration from initiation of zanubrutinib maintenance therapy to disease progression, CR recurrence, or death, whichever occurred first.
Overall survival (OS) | up to 36 months
  OS was defined as the duration from the date of initiation of zanubrutinib maintenance therapy to the date of death.
adverse event | Adverse events were assessed during 3, 6, and 12 months after the start of zanubrutinib maintenance therapy and 6, 12, and 24 months after the end of treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Bei Liu, MD, Principal Investigator — The First Hospital of Lanzhou University,Lanzhou,Gansu,China
Locations (1):
- The First Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
After the completion of the clinical trial, we will choose whether to disclose the result according to the relevant regulations of the Chinese Genetic Office.

REFERENCES:
- [Background] Maurer MJ, Ghesquieres H, Jais JP, Witzig TE, Haioun C, Thompson CA, Delarue R, Micallef IN, Peyrade F, Macon WR, Jo Molina T, Ketterer N, Syrbu SI, Fitoussi O, Kurtin PJ, Allmer C, Nicolas-Virelizier E, Slager SL, Habermann TM, Link BK, Salles G, Tilly H, Cerhan JR. Event-free survival at 24 months is a robust end point for disease-related outcome in diffuse large B-cell lymphoma treated with immunochemotherapy. J Clin Oncol. 2014 Apr 1;32(10):1066-73. doi: 10.1200/JCO.2013.51.5866. Epub 2014 Feb 18. PMID 24550425
- [Background] Yuan T, Zhang F, Yao Q, Liu Y, Zhu X, Chen P. Maintenance therapy for untreated diffuse large B-cell lymphoma: a systematic review and network meta-analysis. Ther Adv Hematol. 2021 May 29;12:20406207211018894. doi: 10.1177/20406207211018894. eCollection 2021. PMID 34104373
- [Background] Pal Singh S, Dammeijer F, Hendriks RW. Role of Bruton's tyrosine kinase in B cells and malignancies. Mol Cancer. 2018 Feb 19;17(1):57. doi: 10.1186/s12943-018-0779-z. PMID 29455639
- [Background] Tam CS, Opat S, D'Sa S, Jurczak W, Lee HP, Cull G, Owen RG, Marlton P, Wahlin BE, Sanz RG, McCarthy H, Mulligan S, Tedeschi A, Castillo JJ, Czyz J, Fernandez de Larrea C, Belada D, Libby E, Matous JV, Motta M, Siddiqi T, Tani M, Trneny M, Minnema MC, Buske C, Leblond V, Trotman J, Chan WY, Schneider J, Ro S, Cohen A, Huang J, Dimopoulos M. A randomized phase 3 trial of zanubrutinib vs ibrutinib in symptomatic Waldenstrom macroglobulinemia: the ASPEN study. Blood. 2020 Oct 29;136(18):2038-2050. doi: 10.1182/blood.2020006844. PMID 32731259
- [Background] Byrd JC, Furman RR, Coutre SE, Burger JA, Blum KA, Coleman M, Wierda WG, Jones JA, Zhao W, Heerema NA, Johnson AJ, Shaw Y, Bilotti E, Zhou C, James DF, O'Brien S. Three-year follow-up of treatment-naive and previously treated patients with CLL and SLL receiving single-agent ibrutinib. Blood. 2015 Apr 16;125(16):2497-506. doi: 10.1182/blood-2014-10-606038. Epub 2015 Feb 19. PMID 25700432
- [Background] Phillips T, Chan H, Tam CS, Tedeschi A, Johnston P, Oh SY, Opat S, Eom HS, Allewelt H, Stern JC, Tan Z, Novotny W, Huang J, Trotman J. Zanubrutinib monotherapy in relapsed/refractory indolent non-Hodgkin lymphoma. Blood Adv. 2022 Jun 14;6(11):3472-3479. doi: 10.1182/bloodadvances.2021006083. PMID 35390135